CLINICAL TRIAL: NCT02592993
Title: Clinical Study to Evaluate the Performance of the PicoWayTM Picosecond Fractional Laser for Treatment of Acne Scars
Brief Title: Performance of PicoWayTM Picosecond Fractional Laser for Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF17261
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PicoWay treatment to all subjects (Experimental): Subjects in this study will receive up to six (6) treatments in 3-8 weeks interval, with the PicoWay device-fractional handpiece 532nm and/or 1064nm according to the study protocol. Subjects will be followed by phone 7 days post first treatment by study staff, and will return for two follow-up (FU) visits at the clinic at: 6 weeks and 12 weeks following the last treatment.
  Interventions: Device: PicoWay device

INTERVENTIONS:
Device: PicoWay device — The PicoWay base unit using a single, free-running, flashlamp-pumped alexandrite laser as a pump source for both the oscillator and the amplifier.

SUMMARY:
Open-label, prospective study. Up to 60 healthy adult volunteers seeking facial acne scars treatment, males or females of 18 to 75 years of age, from up to 3 investigational sites.

DETAILED DESCRIPTION:
Subjects in this study will receive up to six (6) treatments in 3-8 weeks interval, with the PicoWayTM device-fractional handpiece 532nm and/or 1064nm according to the study protocol. Subjects will be followed by phone 7 days post first treatment by study staff, and will return for two follow-up (FU) visits at the clinic at: 6 weeks and 12 weeks following the last treatment.

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 75 years of age
2. Has Fitzpatrick skin type I-VI
3. Subjects seeking treatment for acne scars and wishes to undergo laser treatments for improvement
4. Have bilateral moderate to severe facial acne scars
5. Willing to receive the proposed PicoWayTM fractional treatments and comply with all study (protocol) requirements
6. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications and presentations (subject identity will be masked)
7. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
8. Informed consent process is completed and subject consent is signed

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Hypersensitivity to light exposure
3. Active sun tan in facial area
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
5. Is taking medication(s) for which sunlight is a contraindication
6. Has a history of squamous cell carcinoma or melanoma
7. History of keloid scarring, abnormal wound healing and / or prone to bruising
8. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
9. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness.
10. A laser procedure, a peel or has used lightening creams that was performed in the area to be treated with the past six months
11. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
12. Known allergy to lidocaine, tetracaine, Xylocaine or epinephrine
13. Subjects with pigmented lesions that are considered not acceptable by the study investigator or any condition that, in the investigator's opinion, would make it unsafe to treat.
14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-05-23 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the PicoWayTM treatment | from day 0 up to 13 months
  assessed by blinded evaluators following 3 or 5 treatments, or at 12 weeks post final treatment.

SECONDARY OUTCOMES:
Safety of the PicoWayTM | from day 0 up to 13 months
  assessed by study investigator during all study visits (treatments and follow-up).
efficacy of the PicoWayTM fractional treatment by the investigator | after 3 weeks up to 13 months
  assessed by study investigator during all study visits (starting from the second treatment).
Evaluate investigator satisfaction post treatments | after 46 weeks and after 52 weeks
  assessed by investigator satisfaction post treatments
subject satisfaction post treatments | after 46 weeks and after 52 weeks
  assessed by subject satisfaction post treatments.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dr. Jerome M. Garden, Chicago, Illinois
  - New York Laser & Skin Care, New York, New York
  - Dr. Eric F. Bernstein, Ardmore, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoang Viet M, Derreumaux P, Li MS, Roland C, Sagui C, Nguyen PH. Picosecond dissociation of amyloid fibrils with infrared laser: A nonequilibrium simulation study. J Chem Phys. 2015 Oct 21;143(15):155101. doi: 10.1063/1.4933207. PMID 26493925